CLINICAL TRIAL: NCT00377416
Title: Preclinical & Phase I/II Trials of AAV-AAT Vectors: Phase I Trial of Intramuscular Injection of a Recombinant Adeno-Associated Virus Alpha 1-Antitrypsin (rAAV2-CB-hAAT) Gene Vector to AAT-Deficient Adults
Brief Title: Experimental Gene Transfer Procedure to Treat Alpha 1-Antitrypsin Deficiency
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Alpha-1 Foundation (Other); University of Florida (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 366; R01HL069877 (NIH); NIH Protocol # 30104-465 (Other: NIH); UF GCRC # 567 (Other: University of Florida); UF IBC RD 2101 (University of Florida); UF GTC TRF AAV001; IRB # 306-03
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Gene Transfer Techniques; Gene Therapy
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): rAAV2-CB-hAAT Gene Vector
  Interventions: Genetic: rAAV2-CB-hAAT Gene Vector

INTERVENTIONS:
Genetic: rAAV2-CB-hAAT Gene Vector — Participants will attend a 5-day inpatient visit, during which they will receive a series of injections consisting of one of four different doses of rAAV2-CB-hAAT.

SUMMARY:
Individuals with a deficiency of the Alpha 1-antitrypsin (AAT) protein are at risk for developing emphysema and liver damage. Researchers have developed a way to introduce normal AAT genes into muscle cells so that the AAT protein is produced at normal levels. This study will evaluate the safety of the experimental gene transfer procedure in individuals with AAT deficiency.

DETAILED DESCRIPTION:
AAT deficiency is a genetic disorder in which individuals have inadequate levels of the AAT protein. AAT protects the lungs from white blood cell enzymes that can damage air sacs within the lungs, potentially leading to emphysema. Experimental gene transfer procedures, in which normal copies of genes are inserted into cells, are being developed to treat many genetic diseases, including AAT deficiency. In this study, a modified virus, adeno-associated virus (AAV), has been genetically engineered to contain a normal copy of the AAT gene. When AAV is combined with the AAT gene, the resulting agent, rAAV2-CB-hAAT, is able to carry normal copies of the AAT gene into muscle cells to produce additional AAT. The purpose of this study is to evaluate the safety of injecting rAAV2-CB-hAAT into individuals with AAT deficiency.

This 13-month study will enroll individuals with AAT deficiency. Participants currently using AAT protein replacement will discontinue its use for 15 weeks during the study. Participants will first attend a baseline study visit, which will include a medical history review; a physical examination; an electrocardiogram (ECG) to record heart activity; blood, urine, and semen collection; pulmonary function tests; and chest and arm scans. Participants will then attend a 5-day inpatient visit, during which they will receive a series of injections consisting of one of four different doses of rAAV2-CB-hAAT. Physical examinations will occur on all 5 inpatient days; pulmonary function testing, arm circumference measurements, and collection of blood, urine, and semen will occur on selected days of the inpatient stay. Follow-up study visits, with possible overnight stays, will occur on Days 14 and 90. On Days 30, 45, 60, 75, 180, 270, and 365, participants will have blood drawn at a local clinic. On these same days, study staff will contact participants by telephone to review their medical history and symptoms. Unused blood and semen samples will be frozen and stored for future research purposes. Participants will have yearly follow-up evaluations by either telephone or mail for a total of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AAT deficiency
* Forced expiratory volume in one second (FEV1) greater than 24% of predicted value (post bronchodilator)
* Willing to discontinue AAT protein replacement 4 weeks prior to study entry, and to resume 11 weeks after rAAV2-CB-hAAT has been administered
* Willing to discontinue aspirin, aspirin-containing products, and other drugs that may alter platelet function 7 days prior to study entry, and to resume 24 hours after rAAV2-CB-hAAT has been administered
* Willing to use contraception throughout the study

Exclusion Criteria:

* Required antibiotic therapy for a respiratory infection in the 28 days prior to rAAV2-CB-hAAT administration
* Required oral or systemic corticosteroids in the 28 days prior to rAAV2-CB-hAAT administration
* Liver disease
* Currently receiving or has received an investigational study agent in the 30 days prior to study entry
* Received gene transfer agents in the 6 months prior to study entry
* Currently smokes cigarettes or uses illegal drugs
* History of immune response to human AAT replacement
* History of platelet dysfunction
* Any other medical condition that the investigator deems unsuitable for study participation
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-03; Primary Completion 2006-10 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Arm circumference | Measured at Day 3
Presence of rAAV2-CB-hAAT vector in blood and semen | Measured at Day 14
Serum chemistries, hematology, urinalysis, immune response, and pulmonary function | Measured at Day 90
Human AAT levels and phenotype in the blood | Measured at Day 180
Adverse events | Measured at Year 1 and at yearly follow-up evaluations over 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Terence R. Flotte, MD, Principal Investigator — UMass Medical School
Locations (2):
- United States (2):
  - University of Florida, College of Medicine, Department of Pediatrics, Gainesville, Florida
  - UMass Medical School, Worcester, Massachusetts

REFERENCES:
- [Background] Flotte TR, Brantly ML, Spencer LT, Byrne BJ, Spencer CT, Baker DJ, Humphries M. Phase I trial of intramuscular injection of a recombinant adeno-associated virus alpha 1-antitrypsin (rAAV2-CB-hAAT) gene vector to AAT-deficient adults. Hum Gene Ther. 2004 Jan;15(1):93-128. doi: 10.1089/10430340460732490. PMID 14965381
- [Background] Song S, Morgan M, Ellis T, Poirier A, Chesnut K, Wang J, Brantly M, Muzyczka N, Byrne BJ, Atkinson M, Flotte TR. Sustained secretion of human alpha-1-antitrypsin from murine muscle transduced with adeno-associated virus vectors. Proc Natl Acad Sci U S A. 1998 Nov 24;95(24):14384-8. doi: 10.1073/pnas.95.24.14384. PMID 9826709
- [Derived] Remih K, Amzou S, Strnad P. Alpha1-antitrypsin deficiency: New therapies on the horizon. Curr Opin Pharmacol. 2021 Aug;59:149-156. doi: 10.1016/j.coph.2021.06.001. Epub 2021 Jul 10. PMID 34256305